CLINICAL TRIAL: NCT03840915
Title: A Phase Ib/II, Open-Label Study of M7824 in Combination With Chemotherapy in Participants With Stage IV Non-small Cell Lung Cancer
Brief Title: M7824 in Combination With Chemotherapy in Stage IV Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0024; 2018-004040-28 (EudraCT Number)
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small Cell Lung Cancer; Bintrafusp alfa (proposed INN); M7824; Stage IV; INTR@PID LUNG 024
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin; Pemetrexed; 130-nm albumin-bound paclitaxel; Gemcitabine; Docetaxel; bintrafusp alfa protein, human; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Cisplatin or Carboplatin + Pemetrexed + Bintrafusp alfa (Experimental): Participants received 2400 miligrams (mg) Bintrafusp alfa along with Cisplatin or Carboplatin, and Pemetrexed every 3 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: M7824
- Cohort B: Carboplatin + Paclitaxel or Nab-paclitaxel + Bintrafusp alfa (Experimental): Participants received 2400 mg Bintrafusp alfa along with Carboplatin, and Paclitaxel or Nab-paclitaxel every 3 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
  Interventions: Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Bintrafusp alfa; Drug: Paclitaxel
- Cohort C: Cisplatin or Carboplatin + Gemcitabine + Bintrafusp alfa (Experimental): Participants received 2400 mg Bintrafusp alfa along with Cisplatin or Carboplatin, and Gemcitabine every 3 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Carboplatin; Drug: Bintrafusp alfa
- Cohort D: Docetaxel + Bintrafusp alfa (Experimental): Participants received 2400 mg Bintrafusp alfa along with Docetaxel every 3 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
  Interventions: Drug: Docetaxel; Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Cisplatin — Cisplatin was administered intravenously at a dose of 75 milligrams per meter square (mg/m^2) over 60 minutes every 21 days for 4 cycles (each cycle is 21 days).
  Arms: Cohort A: Cisplatin or Carboplatin + Pemetrexed + Bintrafusp alfa; Cohort C: Cisplatin or Carboplatin + Gemcitabine + Bintrafusp alfa
Drug: Carboplatin — Carboplatin was administered at area under the concentration-time Curve (AUC) 5 when combined with pemetrexed over 30 to 60 minutes every 21 days for 4 cycles (each cycle is 21 days).
  Arms: Cohort A: Cisplatin or Carboplatin + Pemetrexed + Bintrafusp alfa
Drug: Pemetrexed — Pemetrexed was administered intravenously at a dose of 500 mg/ m^2 over 10 minutes every 21 days.
  Arms: Cohort A: Cisplatin or Carboplatin + Pemetrexed + Bintrafusp alfa
Drug: Nab-paclitaxel — Nab-paclitaxel was administered intravenously at as dose of 100 mg/m^2 over 30 minutes in a 21 days cycle on Day 1, 8, and 15 in each cycle for 4 cycles (each cycle is 21 days).
  Arms: Cohort B: Carboplatin + Paclitaxel or Nab-paclitaxel + Bintrafusp alfa
Drug: Gemcitabine — Gemcitabine was administered intravenously at a dose of 1250 mg/m^2 over 30 minutes in a 21 days cycle on Day 1, and 8, in each cycle for 4 cycles (each cycle is 21 days).
  Arms: Cohort C: Cisplatin or Carboplatin + Gemcitabine + Bintrafusp alfa
Drug: Docetaxel — Docetaxel was administered intravenously at a dose of 75 mg/m^2 over 60 minutes every 21 days for 4 cycles (each cycle is 21 days).
  Arms: Cohort D: Docetaxel + Bintrafusp alfa
Drug: M7824 — M7824 was administered intravenously at a dose of 2400 mg every 21 days in combination with chemotherapy for 4 cycles (each cycle is 21 days) followed by up to 31 cycles in maintenance with M7824 and pemetrexed.
  Arms: Cohort A: Cisplatin or Carboplatin + Pemetrexed + Bintrafusp alfa
Drug: Carboplatin — Carboplatin was administered at area under the concentration-time Curve (AUC) 6 when combined with nab-paclitaxel over 30 to 60 minutes every 21 days for 4 cycles (each cycle is 21 days).
  Arms: Cohort B: Carboplatin + Paclitaxel or Nab-paclitaxel + Bintrafusp alfa
Drug: Carboplatin — Carboplatin was administered at area under the concentration-time Curve (AUC) 5 when combined with gemcitabine over 30 to 60 minutes every 21 days for 4 cycles (each cycle is 21 days).
  Arms: Cohort C: Cisplatin or Carboplatin + Gemcitabine + Bintrafusp alfa
Drug: Bintrafusp alfa — M7824 was administered intravenously at a dose of 2400 mg every 21 days in combination with chemotherapy for 4 cycles (each cycle is 21 days) followed by up to 31 cycles in maintenance with M7824 alone.
  Arms: Cohort B: Carboplatin + Paclitaxel or Nab-paclitaxel + Bintrafusp alfa; Cohort C: Cisplatin or Carboplatin + Gemcitabine + Bintrafusp alfa; Cohort D: Docetaxel + Bintrafusp alfa
Drug: Paclitaxel — Paclitaxel was administered intravenously at a dose of 200 mg/m2 over 3 hours every 3 weeks for 4 cycles (each cycle is 21 days).
  Arms: Cohort B: Carboplatin + Paclitaxel or Nab-paclitaxel + Bintrafusp alfa

SUMMARY:
The main purpose of the study was to evaluate the safety and tolerability of M7824 in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants greater than or equals to (>=) 18 years of age inclusive at the time of signing the informed consent
* Participants who have histologically confirmed diagnosis of Stage IV NSCLC:

  1. Participants in Cohort A, B, and C must not have received prior systemic therapy treatment for their Stage IV NSCLC
  2. Participants who had disease progression on previous treatment with Programmed death-ligand 1 (PD- L1) inhibitors in combination with platinum-based chemotherapy are enrolled in Cohort D, as long as therapy was completed at least 28 days of the first study intervention.
* Have measurable disease based on Response evaluation criteria in solid tumors (RECIST) 1.1
* Have a life expectancy of at least 3 months
* Availability of archived tumor material (less than [<] 6 months old) adequate for biomarker analysis is mandatory at Screening, central laboratory confirmation is required. Fresh biopsies should be collected if archived tumor material is not available
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at study entry and date of first dose

Exclusion Criteria:

* The participant's tumor harbors an epidermal growth factor receptor (EGFR) sensitizing (activating) mutation,ROS1 rearrangement, or BRAF V600E mutation or anaplastic lymphoma kinase (ALK) positive, if targeted therapy is locally approved
* Mixed small cell with NSCLC cancer histology
* Has received major surgery within 4 weeks prior to the first dose of study intervention; received thoracic radiation therapy (RT) of > 30 gray (Gy) within 6 months prior to the first dose of study intervention
* Previous malignant disease (other than the target malignancy to be investigated in this study) within the last 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are clinically stable for at least 2 weeks after the end of the RT and, have no evidence of new or enlarging brain metastases evaluated by imaging, preferably brain magnetic resonance imaging (MRI)
* Known severe hypersensitivity to study intervention or any components in their formulations
* For participants in Cohort A, B and C: Has received prior systemic therapy for Stage IV NSCLC, including anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Unable to tolerate computed tomography (CT) or MRI in the opinion of the Investigator and/or allergy to contrast material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (19):
- United States (8):
  - Compassionate Care Research Group Inc - Edinger Medical Group, Inc., Fountain Valley, California
  - California Cancer Associates for Research & Excellence, Inc., San Marcos, California
  - Hematology - Oncology Associates of Treasure Coast - Hematology-Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Baptist Health Lexington Oncology Associates, Lexington, Kentucky
  - University of Maryland - DUPLICATE/Pediatric Surgery, Baltimore, Maryland
  - RCCA MD LLC - Bethesda, Bethesda, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Belgium (5):
  - Universitair Ziekenhuis Brussel - Geriatrie, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent - Medical Oncology, Ghent
  - CHU Sart Tilman, Liège
  - AZ Sint-Maarten, Mechelen
- France (6):
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Maison du Ha, Bordeaux
  - Centre Georges François Leclerc - Unité de Phase I, Dijon
  - Hôpital de la Timone# - CPCEM CIC - Bat F 1er étage, Marseille
  - ICO - Site René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Poitiers - Hôpital la Milétrie - service d'oncologie médicale, Poitiers

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] Vugmeyster Y, Grisic AM, Wilkins JJ, Loos AH, Hallwachs R, Osada M, Venkatakrishnan K, Khandelwal A. Model-informed approach for risk management of bleeding toxicities for bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1. Cancer Chemother Pharmacol. 2022 Oct;90(4):369-379. doi: 10.1007/s00280-022-04468-6. Epub 2022 Sep 6. PMID 36066618
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0024
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 127 participants were screened out of which 70 participants who received study intervention.
Groups:
- Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed: Participants received 2400 miligrams (mg) Bintrafusp alfa along with Cisplatin 75 mg/ m^2 (per meter square) over 60 minutes or Carboplatin at area under the concentration-time Curve (AUC) 5 when combined with pemetrexed at a dose of 500 mg/ m^2 over 30 to 60 minutes every 21 days for 4 cycles (each cycle is 21 days) until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
- Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel: Participants received 2400 mg Bintrafusp alfa along with Carboplatin at area under the concentration-time Curve (AUC) 6 when combined with nab-paclitaxel at as dose of 100 mg/m^2 over 30 to 60 minutes(Nab- paclitaxel was administered on Day 1, 8, and 15), and Paclitaxel at a dose of 200 mg/m2 over 3 hours every 21 days for 4 cycles until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
- Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine: Participants received 2400 mg Bintrafusp alfa along with Cisplatin at a dose of 75 milligrams per meter square (mg/m^2) over 60 minutes or Carboplatin at area under the concentration-time Curve (AUC) 5 when combined with gemcitabine at a dose of 1250 mg/m^2 over 30 to 60 minutes every 21 days for 4 cycles until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
- Cohort D: Bintrafusp Alfa + Docetaxel: Participants received 2400 mg Bintrafusp alfa along with Docetaxel at a dose of 75 mg/m^2 over 60 minutes every 21 days for 4 cycles until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
Period: Overall Study
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Started | 40 | 9 | 9 | 12
Safety Analysis Set (All participants who were administered any dose of any study intervention (bintrafusp alfa or one of the chemotherapies).) | 40 | 9 | 9 | 12
Full Analysis Set (All participants who were administered any dose of any study intervention (bintrafusp alfa or one of the chemotherapies).) | 40 | 9 | 9 | 12
Dose-Limiting Toxicity Analysis Set (All participants who received at least 90% of the bintrafusp alfa infusion and all other planned study administrations during the DLT observation period of 3 weeks and who did not discontinue the study for other reasons than DLT during the first cycle, or who experienced at least one DLT.) | 8 | 8 | 8 | 11
Completed | 40 | 9 | 9 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel | Total
Number analyzed (Participants) | 40 | 9 | 9 | 12 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (10.3) | 64 (8.7) | 61 (11.2) | 60 (7.7) | 62 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 4 | 7 | 23
  Male | 31 | 6 | 5 | 5 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity-Not Hispanic or Latino | 15 | 8 | 3 | 3 | 29
  Ethnicity-Unknown or Not Reported | 25 | 1 | 6 | 9 | 41
  Race-Black or African American | 1 | 2 | 0 | 0 | 3
  Race-White | 14 | 6 | 2 | 3 | 25
  Race-Other | 0 | 0 | 1 | 0 | 1
  Race-Not Collected | 25 | 1 | 6 | 9 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as Adverse Events(AEs) with any of following toxicities: Grade 4 nonhematologic toxicity or hematologic toxicity lasting more than equal to(>=) 7 days despite medical intervention; Grade 3 nausea, vomiting, and diarrhea lasting >= 3 days despite supportive care; Any Grade 3 or Grade 4 nonhematologic lab value leading to hospitalization or persisting for >= 7 days; Grade 3 or Grade 4: grade 3 is defined as absolute neutrophil count (ANC) less than (<) 1,000/Cubic Millimeter(mm3) with a temperature of > 38.3 degree Celsius (°C); grade 4 is defined as ANC < 1,000/mm3 with a temperature of > 38.3°C, with life-threatening consequences; Thrombocytopenia < 25,000/mm3 associated with bleeding not resulting in hemodynamic instability or a life-threatening bleeding resulting in urgent intervention; Bleeding events >= Grade 3 occurring within 5 days of bintrafusp alfa treatment; Prolonged delay(> 3 weeks) in initiating Cycle 2 due to treatment-related toxicity; Grade 5 toxicity.
Time Frame: Day 1 Week 1 up to Week 3
Population: Dose-Limiting Toxicity Analysis (DLT) Set included all participants who received at least 90 percent (%) of the bintrafusp alfa infusion and all other planned study administrations during the DLT observation period of 3 weeks and who did not discontinue the study for other reasons than DLT during the first cycle, or who experienced at least one DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 8 | 8 | 8 | 11
Participants | 1 | 1 | 0 | 3

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether considered related to the medicinal product or protocol-specified procedure. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAE was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious TEAEs and non-serious TEAEs.
Time Frame: Time from first treatment assessed up to approximately 26 months
Population: The safety analysis set (SAF) included all participants who were administered any dose of any study intervention (bintrafusp alfa or one of the chemotherapies).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 40 | 9 | 9 | 12
Participants
  TEAEs | 40 | 9 | 9 | 12
  Serious TEAEs | 31 | 5 | 6 | 9

3. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator (IRC)
Description: Percentage of participants with confirmed objective response that is at least one overall assessment of complete response (CR) or partial response (PR) reported here. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by Investigator.
Time Frame: Time from first treatment assessed up to approximately 26 months
Population: The full analysis set (FAS) included all participants who were administered any dose of any study intervention (bintrafusp alfa or one of the chemotherapies).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 40 | 9 | 9 | 12
Percentage of Participants | 45.0 [29.3 to 61.5] | 66.7 [29.9 to 92.5] | 44.4 [13.7 to 78.8] | 16.7 [2.1 to 48.4]

4. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Investigator
Description: PFS was defined as the time from first administration of study intervention until date of the first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Kaplan-Meier estimates was used to calculate PFS.
Time Frame: Time from first administration of study drug until the first documentation of PD or death, assessed up to approximately 26 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 40 | 9 | 9 | 12
months | 5.0 [0.0 to 14.3] | 4.1 [1.2 to 17.7] | 5.4 [1.4 to 19.6] | 2.6 [1.3 to 10.4]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first administration of study intervention to the date of death due to any cause. The OS was analyzed by using the Kaplan-Meier method.
Time Frame: Time from first treatment assessed up to approximately 26 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 40 | 9 | 9 | 12
months | 11.4 [6.4 to 15.1] | 11.8 [1.9 to NA] — Due to small number of events, estimate (upper limit of 95% confidence interval) from Kaplan-Meier survival curves could not be derived. | NA [5.7 to NA] — Due to small number of events, estimate (Median and upper limit of 95% confidence interval) from Kaplan-Meier survival curves could not be derived. | 16.5 [3.0 to NA] — Due to small number of events, estimate (upper limit of 95% confidence interval) from Kaplan-Meier survival curves could not be derived.

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined for participants with confirmed response, as the time from first documentation of confirmed objective response (Complete Response [CR] or Partial Response [PR]) according to RECIST 1.1 to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Results were calculated based on Kaplan-Meier estimates.
Time Frame: Time from first documentation of a confirmed objective response to PD or death due to any cause (assessed up to approximately 26 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 40 | 9 | 9 | 12
months | 9.6 [3.7 to NA] — Due to small number of events, estimate (upper limit of 95% confidence interval) from Kaplan-Meier survival curves could not be derived. | NA [2.8 to NA] — Due to small number of events, estimate (Median and upper limit of 95% confidence interval) from Kaplan-Meier survival curves could not be derived. | 10.5 [2.8 to NA] — Due to small number of events, estimate (upper limit of 95% confidence interval) from Kaplan-Meier survival curves could not be derived. | 3.4 [3.0 to 3.8]

7. Secondary Outcome: Immediate Observed Serum Concentration at End of Infusion (Ceoi) of Bintrafusp Alfa
Description: Ceoi was the observed concentration at the end of the infusion period. This was taken directly from the observed Bintrafusp Alfa concentration-time data.
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: In the context of Study NCT03631706, NCT04066491, and NCT03840902 been terminated prematurely, the sponsor decided to restrict the analyses of Pharmacokinetics (PK) Parameter and no PK data was collected.
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Serum Trough Concentration Levels (Ctrough) of Bintrafusp Alfa
Description: Ctrough was the serum concentration observed immediately before next dosing.
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: as for outcome 7
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Bintrafusp Alfa
Description: The area under the concentration-time curve (AUC) from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: as for outcome 7
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Bintrafusp Alfa
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from terminal first order (elimination) rate constant determination. AUC0-inf= AUC0-tlast +Clast pred/ terminal first order (elimination) rate constant.
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: as for outcome 7
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bintrafusp Alfa
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: as for outcome 7
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Bintrafusp Alfa
Description: The time to reach the maximum observed concentration collected during a dosing interval. Tmax was obtained directly from the concentration versus time curve.
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: as for outcome 7
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Bintrafusp Alfa
Description: Elimination half-life determined as 0.693/terminal first order (elimination) rate constant.
Time Frame: Predose, Day 22, Day 43, Day 64 and Day 85
Population: as for outcome 7
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADA)
Description: Serum samples were analyzed by a validated assay method to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: Time from first treatment assessed up to approximately 26 months
Population: Immunogenicity Analysis Set included all participants who have received at least of 1 dose of bintrafusp alfa + chemotherapy and had at least 1 valid antidrug antibody result.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
Number analyzed (Participants) | 38 | 9 | 8 | 12
Participants | 9 | 3 | 2 | 3

ADVERSE EVENTS:
Time Frame: Time from first treatment assessed up to approximately 26 months
Arm/Group | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine | Cohort D: Bintrafusp Alfa + Docetaxel
All-Cause Mortality (participants affected / at risk) | 23/40 | 4/9 | 4/9 | 6/12
Serious Adverse Events (participants affected / at risk) | 31/40 | 5/9 | 6/9 | 9/12
Other Adverse Events (participants affected / at risk) | 40/40 | 9/9 | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed (N=40) | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel (N=9) | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine (N=9) | Cohort D: Bintrafusp Alfa + Docetaxel (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (4) | 0 (0) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophilus sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yersinia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Bintrafusp Alfa + Cisplatin/Carboplatin + Pemetrexed (N=40) | Cohort B: Bintrafusp Alfa + Carboplatin + Paclitaxel or Nab-paclitaxel (N=9) | Cohort C: Bintrafusp Alfa + Cisplatin/Carboplatin + Gemcitabine (N=9) | Cohort D: Bintrafusp Alfa + Docetaxel (N=12)
Anaemia (Blood and lymphatic system disorders) | 20 (28) | 6 (12) | 9 (9) | 9 (9)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (5) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 1 (3) | 5 (5) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (13) | 2 (3) | 4 (6) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (10) | 6 (10) | 2 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 13 (15) | 3 (3) | 2 (2) | 6 (10)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (29) | 3 (3) | 6 (11) | 5 (5)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosa erosion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 2 (6) | 0 (0) | 2 (2)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (12) | 1 (1) | 2 (4) | 5 (6)
Asthenia (General disorders) | 15 (20) | 1 (1) | 4 (10) | 7 (10)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Chills (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 7 (9) | 3 (3) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 6 (8) | 0 (0) | 2 (3) | 3 (3)
Pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 11 (16) | 1 (1) | 0 (0) | 4 (6)
Xerosis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yersinia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 3 (5) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 0 (0) | 2 (3) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 1 (4) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0) | 3 (6) | 2 (2)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Gastric pH decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (7) | 3 (5) | 1 (3) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (6) | 0 (0) | 2 (5) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (9) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (12) | 4 (6) | 1 (3) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9) | 3 (4) | 4 (4) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (2) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (9) | 3 (6) | 1 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (5) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (11) | 4 (15) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 1 (1) | 1 (1) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Pica (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4) | 1 (1) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 1 (1) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 1 (1) | 4 (6) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 2 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 2 (8) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0) | 2 (2) | 2 (3)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (22) | 3 (3) | 6 (11) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (2) | 2 (3) | 2 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (6) | 1 (12) | 0 (0)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Artery dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 7 (8) | 3 (3) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03840915/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT03840915/SAP_001.pdf